CLINICAL TRIAL: NCT02991027
Title: OCT Image Quality Performance Evaluation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects needed for enrollment anymore
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Topcon Tabil-801-2016
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-10

CONDITIONS: Healthy Eyes
Keywords: no known ocular pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects Presenting With Normal Eyes (Experimental): Subjects with no known ocular diseases will be imaged using 2 different light sources using the DRI Triton
  Interventions: Device: DRI OCT Triton

INTERVENTIONS:
Device: DRI OCT Triton — DRI OCT Triton using micro-electro-mechanical short cavity tunable laser
Device: DRI OCT Triton — DRI OCT Triton using micro-electro-mechanical tunable vertical cavity surface emitting laser

SUMMARY:
To evaluate the image qualities and segmentation performance of Topcon's DRI OCT Triton devices using two light sources.

DETAILED DESCRIPTION:
To evaluate the image qualities and segmentation performance of Topcon's DRI OCT Triton devices using two light sources with equivalent specifications: the micro-electro-mechanical short cavity tunable laser and the micro-electro-mechanical tunable vertical cavity surface emitting laser.

ELIGIBILITY:
Inclusion Criteria

1. Participants must be at least 18 years of age
2. They must be able to complete all testing (all OCT scans)
3. They must volunteer to be in the study and sign the consent form

Exclusion Criteria

1. Subject with history of ocular disease or ocular pathology
2. Subjects unable to complete all OCT imaging modes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
OCT image quality | 5 minutes
OCT angiography image quality | 5 minutes

SECONDARY OUTCOMES:
Full Retinal Thickness | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Wang, PhD, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon Medical Systems Inc., Oakland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No